CLINICAL TRIAL: NCT06931665
Title: Neurological and Physiological Effects of Animal-assisted Therapy for Patients in a Minimally Conscious State: a Randomized, Controlled Cross-over Study
Brief Title: Neurological and Physiological Effects of Animal-assisted Therapy for Patients in a Minimally Conscious State
Acronym: EMCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: Rehab Basel (Other)
Responsible Party: Principal Investigator, Fabio Carbone, Doctoral Assistant, University of Basel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02318; PCEFP1_194591 / 1 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2025-03-26; First posted 2025-04-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Minimally Conscious State
MeSH Terms: conditions — Persistent Vegetative State | interventions — Animal Assisted Therapy; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, controlled cross-over within-subject trial with two arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAT-TAU-AAT-TAU (arm 1) (Experimental): Each patient will undergo two therapy sessions per week, with a total of four sessions integrated into their clinical routine. In this arm, patients will start with the AAT intervention, followed by a TAU intervention in the same week. In week two, the patient will again receive an AAT intervention followed by the last TAU intervention.
  Interventions: Procedure: Animal Assisted Occupational Therapy
- TAU-AAT-TAU-AAT (arm 2) (Experimental): Each patient will undergo two therapy sessions per week, with a total of four sessions integrated into their clinical routine. In this arm, patients will start with the TAU intervention, followed by an AAT intervention in the same week. In week two, the patient will again receive a TAU intervention followed by the last AAT intervention.
  Interventions: Procedure: Animal Assisted Occupational Therapy

INTERVENTIONS:
Procedure: Animal Assisted Occupational Therapy — AAT is an ergotherapy including an animal. AAT is a specific type of Animal Assisted Intervention (AAI) with a therapeutic aim.
  Other Names: Animal Assisted Therapy; AAT; ergotherapy

SUMMARY:
This study aims to explore the impact of Animal Assisted Therapy (AAT) on brain signal complexity in patients with minimally conscious state (MCS) by analyzing electroencephalogram (EEG) entropy. MCS patients typically exhibit reduced brain entropy compared to healthy individuals, indicating lower brain complexity. The study will assess whether AAT can enhance this complexity, which is crucial for understanding consciousness levels. Entropy, a measure of randomness in brain activity, will be used to evaluate AAT's effectiveness. In addition, electrocardiography (ECG), electrodermal activity (EDA) and behavioral measurements will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients in one of the study sites
* Acquired brain injury resulting from either traumatic or non-traumatic events
* Diagnosis of MCS defined by CRS-R according to the Aspen criteria (Giacino, 2005)
* Informed consent as documented by signature by the patient's legal representative
* Physiologically stable
* Aged 18 or over

Exclusion Criteria:

* Phobia or allergies to any of the involved animals
* Medical contraindications: acute or chronic disease (e.g. chronic pain, hypertension, heart disease, renal disease, liver disease, diabetes)
* Radical changes in medication (decision made with responsible physician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
EEG signal complexity 1 | Before, during and after AAT and TAU. Approximately three weeks.
  The EEG signal complexity is measured via entropy computed based on EEG recordings:
  • Sample Entropy (SampEn): score usually between 0 and 1 with higher score indicating higher entropy
EEG signal complexity 2 | Before, during and after AAT and TAU. Approximately three weeks.
  The EEG signal complexity is measured via entropy computed based on EEG recordings:
  • Lempel-Ziv complexity (LCZ): score usually between 0 and 1 with higher score indicating higher entropy
EEG signal complexity 3 | Before, during and after AAT and TAU. Approximately three weeks.
  The EEG signal complexity is measured via three measures of entropy computed based on EEG recordings:
  • Symbolic Transfer Entropy (STE): score usually between 0 and 1 with higher score indicating higher entropy

SECONDARY OUTCOMES:
Other physiological measures 1 | Before, during and after AAT and TAU. Approximately three weeks.
  • Heart rate (HR) in bpm
Other physiological measures 2 | Before, during and after AAT and TAU. Approximately three weeks.
  • Heart rate variability (HRV) measured by complexity index (CI): score usually between 0 and 1 with higher score indicating higher complexity
Other physiological measures 3 | Before, during and after AAT and TAU. Approximately three weeks.
  • Electrodermal activity (EDA) in uS

OTHER OUTCOMES:
Behavioral data assessing state of consciousness 1 | From enrollment to the end of treatment at 2 weeks. Day 1 and last day
  • Coma Recovery Scale - Revised (CRS-R): score from 0 to 23 with higher score indicating higher consciousness level
Behavioral data assessing state of consciousness 2 | From enrollment to the end of treatment at 2 weeks. Two pre-session measures per week, two post-session measures per week
  • Basler Vegetative State Assessment (BAVESTA): 22 items with a score from 0 to 5 with higher total score indicating higher level of consciousness

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - REHAB Basel, Basel
  - Service de Neurorééducation, Hopitaux Universitaires Genevois, Geneva

IPD SHARING:
Plan to Share IPD: No